CLINICAL TRIAL: NCT06718335
Title: Prospective, Multi-cohort, Exploratory Clinical Study of Pyrrotinib Maleate in HER2-positive Early Breast Cancer
Brief Title: Pyrotinib in HER2-positive Early Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nie Jianyun (Other)
Responsible Party: Sponsor-Investigator, Nie Jianyun, Nie jianyun,MD, Yunnan Cancer Hospital
Organization: Yunnan Cancer Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-YUNNAN-001
Record Dates: First submitted 2024-10-14; First posted 2024-12-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pyrotinib (Experimental): Patients who meet the screening criteria will receive pyrotinib (400mg, qd) + trastuzumab injection (first dose 8mg/kg, subsequent 6mg/kg, d1) + albumin purpurenin (125mg/m2, d1, d8) + carboplatin (AUC=6, d1) for 21 days/cycle for a total of 6 cycles of neoadjuvant therapy. One month after the end of neoadjuvant therapy, patients should receive radical mastectomy (breast-conserving surgery or total mastectomy), if the postoperative pathological complete response patients receive pyrotinib (400mg, qd) for one year,. If patients were hormone receptor positive patients at the adjuvant treatment stage, the endocrine treatment regimen was selected by the investigators.
  Interventions: Drug: Pyrotinib
- T-DM1 (Experimental): Patients who meet the screening criteria will receive pyrotinib (400mg, qd) + trastuzumab injection (first dose 8mg/kg, subsequent 6mg/kg, d1) + albumin purpurenin (125mg/m2, d1, d8) + carboplatin (AUC=6, d1) for 21 days/cycle for a total of 6 cycles of neoadjuvant therapy. One month after the end of neoadjuvant therapy, patients should receive radical mastectomy (breast-conserving surgery or total mastectomy), if the postoperative non-pathological complete response patients with RCB-1 receive Trastuzumab Emtansine (3.6 mg/kg, iv) for one year. If patients were hormone receptor positive patients at the adjuvant treatment stage, the endocrine treatment regimen was selected by the investigators.
  Interventions: Drug: Pyrotinib
- T-DM1 and pertuzumab (Experimental): Patients who meet the screening criteria will receive pyrotinib (400mg, qd) + trastuzumab injection (first dose 8mg/kg, subsequent 6mg/kg, d1) + albumin purpurenin (125mg/m2, d1, d8) + carboplatin (AUC=6, d1) for 21 days/cycle for a total of 6 cycles of neoadjuvant therapy. One month after the end of neoadjuvant therapy, patients should receive radical mastectomy (breast-conserving surgery or total mastectomy), if the postoperative non-pathological complete response patients with RCB≥2 were treated with Trastuzumab Emtansine (3.6 mg/kg, iv) combined with pertuzumab for one year. If patients were hormone receptor positive patients at the adjuvant treatment stage, the endocrine treatment regimen was selected by the investigators.
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Patients who meet the screening criteria will receive pyrotinib (400mg, qd) + trastuzumab injection (first dose 8mg/kg, subsequent 6mg/kg, d1) + albumin purpurenin.In adjuvant therapy, pathological complete response patients receive pyrotinib time to one year, non-pathological complete response patients with RCB-1 receive Trastuzumab Emtansine time to one year，RCB≥2 were treated with Trastuzumab Emtansine combined with pertuzumab time to one year.

SUMMARY:
This is a Multi-cohort, Phase II Clinical Study of Neoadjuvant - Adjuvant Pyrotinib in the Treatment of HER2-positive Early Breast Cancer, To evaluate the efficacy and safety of the pyrotinib-containing study regimen in patients with early HER2-positive early breast cancer with neoadjuvant and postoperative different Residual tumor burden (RCB) scores.

DETAILED DESCRIPTION:
This is a Multi-cohort, Phase II Clinical Study of Neoadjuvant - Adjuvant Pyrotinib in the Treatment of HER2-positive Early Breast Cancer, To evaluate the efficacy and safety of the pyrotinib-containing study regimen in patients with early HER2-positive early breast cancer with neoadjuvant and postoperative different Residual tumor burden scores.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥18 years and ≤75 years with newly treated breast cancer;
2. Pathological examination confirmed HER2 positive (immunohistochemistry staining +++ or immunohistochemistry staining ++ and Fluorescence in situ hybridization positive);
3. Patients with invasive breast cancer diagnosed histologically plus imaging as early (T1c-3, N0-1, M0) or locally advanced (T2-3, N2, or N3, M0);
4. Eastern Cooperative Oncology Group score 0~1;
5. Plan to undergo the final surgical removal of breast cancer, i.e. breast conserving surgery or total mastectomy, sentinel lymph node (SN) biopsy or axillary lymph node dissection (ALND);
6. If the major organs function normally, the following criteria are met:

(1) The standard of blood routine examination should meet: absolute neutrophil count(ANC) ≥1.5×109/L; blood platelet (PLT) ≥90×109/L; Hb ≥90g/L; (2) Biochemical examination should meet the following criteria: total bilirubin(TBIL)≤ upper limit of normal value (ULN); alanine aminotransferase(ALT) and AST≤1.5 times the upper limit of normal (ULN); Alkaline phosphatase ≤2.5 times the upper limit of normal (ULN); blood urea nitrogen(BUN)and Cr≤1.5×ULN and creatinine clearance ≥50 mL/min (CockcroftGault formula); (3) Color Doppler ultrasonography and echocardiography: left ventricular ejection fraction (LVEF≥55%); (4) Fridericia calibrated QT interval (QTcF) for 18-lead ECG <470 ms; 7. For female patients who are not menopausal or have not been surgically sterilized: consent to abstinence or use of an effective contraceptive method during treatment and for at least 7 months after the last dose in the study treatment; 8. Volunteer to join the study and sign the informed consent.

Exclusion Criteria:

1. Known allergic history of the drug components of this protocol;
2. Previously received antitumor therapy or radiation therapy for any malignant tumor (except for cured cervical carcinoma in situ and basal cell carcinoma);
3. Has undergone major non-breast cancer related surgery within 4 weeks, or has not fully recovered from such surgery;
4. Stage IV (metastatic) breast cancer patients;
5. Inability to swallow, intestinal obstruction, or other factors affecting the administration and absorption of the drug;
6. Serious heart disease or discomfort that cannot be treated;
7. Suffering from mental illness or psychotropic substance abuse, unable to cooperate;
8. Pregnant or lactating women;
9. Patients with severe liver and kidney function diseases and blood system diseases;
10. Those who were not considered suitable for inclusion by the researchers included: history of drug abuse, history of use of blood products, anticoagulant drugs and immunological drugs within the past year; Patients with poor compliance and refusal to cooperate with treatment; Patients with severe high blood pressure, diabetes and other doctors deemed unsuitable for joining the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival(EFS) | 3 year
  Event Free Survival

SECONDARY OUTCOMES:
total pathological complete response(tpCR) | 24 month
  total pathological complete response